CLINICAL TRIAL: NCT04628104
Title: CMR Findings in COVID-19 Patients Presenting With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdallah Hamada, principal investigator, Assiut University
Other Study IDs: CMR in myocardial infarction
Record Dates: First submitted 2020-11-12; First posted 2020-11-13 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days

GROUPS / COHORTS (2):
- COVID-19 patients presented with myocardial infarction
  Interventions: Radiation: cardiac magnetic resonance
- Non-COVID-19 patients presented with myocardial infarction
  Interventions: Radiation: cardiac magnetic resonance

INTERVENTIONS:
Radiation: cardiac magnetic resonance — o CMR protocol:
  * Cine imaging to assess regional & global ventricular function according to the AHA 16-segment model.
  * T2-weighted imaging to detect extent & distribution of myocardial edema.
  * Early Gd enhancement imaging to detect extent & distribution of myocardial hyperemia.
  * Late Gd enhancement imaging to detect extent & distribution of myocardial necrosis.
  * Single-short sequences & other acceleration techniques will be used as appropriate in patients with poor ability to hold their breath.
  * Post-processing analysis will be done on a dedicated workstation

SUMMARY:
To compare myocardial injury in COVID 19 patients presented with myocardial infarction and non COVID Patients presented with myocardial infarction evaluated with CMR

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a global pandemic affecting 185 countries and >3 000 000 patients worldwide as of April 28, 2020. COVID-19 is caused by severe acute respiratory syndrome coronavirus 2,. Among patients with COVID-19, there is a high prevalence of cardiovascular disease, and >7% of patients experience myocardial injury from the infection (22% of critically ill patients). Although angiotensin-converting enzyme 2 serves as the portal for infection, the role of angiotensin-converting enzyme inhibitors or angiotensin receptor blockers requires further investigation.

However, much like any other respiratory tract infection, pre-existing cardiovascular disease (CVD) and CV risk factors enhance vulnerability to COVID-19. Further, COVID-19 can worsen underly- ing CVD and even precipitate de novo cardiac complications.

Preliminary reports suggest that haemostatic abnormalities, including disseminated intravascular coagulation (DIC), occur in patients affected by COVID-19. Additionally, the severe inflammatory response, critical illness, and underlying traditional risk factors may all predispose to thrombotic events, similar to prior virulent zoonotic coronavirus outbreaks CMR is the reference non-invasive standard for cardiac function and tissue characterization and may offer an effective and efficient diagnostic imaging choice to obtain critical information for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with symptoms and ECG indicative of acute MI (both STEMI & NSTEMI) AND confirmed COVID-19.
2. Patients admitted with acute MI (both STEMI & NSTEMI) who develop COVID-19 symptoms during hospital admission & are confirmed by RT-PCR to have COVID-19

Exclusion Criteria:

1. History of previous diagnosis of STEMI or myocarditis.
2. History of previous PCI in infarcted related artery or NSTEMI
3. Severe respiratory distress that precludes lying supine in the CMR scanner.
4. Acute kidney injury with rapidly declining GFR or GFR that is persistently below 30 ml/min/1.73 m2 (contraindication for Gadopentetate dimeglumine contrast).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included patients will be randomly divided in a 1:1 pattern into two groups. The 1st group are COVID 19 patients and the 2nd group are non COVID 19 patients as a control.
  All patients will be subjected to:
  A. Full history taking: including age, sex, history of DM, HTN, Smoking, dyslipidemia, symptoms of COVID 19 infection, chest pain analysis.
  B. Thorough physical examination:
  * General examination including Systolic and diastolic blood pressure, heart rate assessment and O2 Saturation
  * Cardiac examination C. Twelve lead ECG: to search for STEMI criteria according to ECS guidelines of STEMI 2017.5 D. lab investigation: Cardiac enzymes, Renal function, Liver function, CBC, CRP, Lipid profile, RBG, Serum ferritin, ESR, D-Dimer, PCR.
  E.MSCT chest: to detect finding suggestive of COVID 19 infection.
  F.CMR:
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
comparison between COVID-19 and COVID-19 presented with myocardial infarction | baseline
  Distribution and Extent of myocardial injury in COVID 19 patients presented with myocardial infarction and non COVID Patients presented with myocardial infarction evaluated with CMR.

CONTACTS AND LOCATIONS:
Locations (1):
- AssuitU, Asyut, Egypt

REFERENCES:
- [Background] Stefanini GG, Montorfano M, Trabattoni D, Andreini D, Ferrante G, Ancona M, Metra M, Curello S, Maffeo D, Pero G, Cacucci M, Assanelli E, Bellini B, Russo F, Ielasi A, Tespili M, Danzi GB, Vandoni P, Bollati M, Barbieri L, Oreglia J, Lettieri C, Cremonesi A, Carugo S, Reimers B, Condorelli G, Chieffo A. ST-Elevation Myocardial Infarction in Patients With COVID-19: Clinical and Angiographic Outcomes. Circulation. 2020 Jun 23;141(25):2113-2116. doi: 10.1161/CIRCULATIONAHA.120.047525. Epub 2020 Apr 30. No abstract available. PMID 32352306
- [Background] Mahmud E, Dauerman HL, Welt FGP, Messenger JC, Rao SV, Grines C, Mattu A, Kirtane AJ, Jauhar R, Meraj P, Rokos IC, Rumsfeld JS, Henry TD. Management of Acute Myocardial Infarction During the COVID-19 Pandemic: A Position Statement From the Society for Cardiovascular Angiography and Interventions (SCAI), the American College of Cardiology (ACC), and the American College of Emergency Physicians (ACEP). J Am Coll Cardiol. 2020 Sep 15;76(11):1375-1384. doi: 10.1016/j.jacc.2020.04.039. Epub 2020 Apr 21. PMID 32330544
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Chen C, Chen C, Yan JT, Zhou N, Zhao JP, Wang DW. [Analysis of myocardial injury in patients with COVID-19 and association between concomitant cardiovascular diseases and severity of COVID-19]. Zhonghua Xin Xue Guan Bing Za Zhi. 2020 Jul 24;48(7):567-571. doi: 10.3760/cma.j.cn112148-20200225-00123. Chinese. PMID 32141280
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967